CLINICAL TRIAL: NCT06273410
Title: Clinical Performance of An Alkasite Based Restorative Material With And Without Adhesive (A Randomized Controlled Clinical Trial)
Brief Title: Clinical Performance of An Alkasite Based Restorative Material With And Without Adhesive
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hams Hamed Abdelrahman (Other)
Responsible Party: Sponsor-Investigator, Hams Hamed Abdelrahman, Assistant lecturer of DPH and Clinical statistician, Alexandria University
Organization: Alexandria University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 0453-6/2022
Record Dates: First submitted 2024-02-02; First posted 2024-02-22 (Actual); Last update posted 2024-02-22 (Actual); Status verified 2024-02

CONDITIONS: Dental Restoration Failure
MeSH Terms: interventions — Adhesives

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cention N without adhesive. (Experimental)
  Interventions: Other: Cention N
- Cention N with adhesive (Experimental)
  Interventions: Other: Cention N + Adhesive
- Filtek Bulk Fill posterior composite (Active Comparator)
  Interventions: Other: Bulk Fill Composite

INTERVENTIONS:
Other: Cention N — Cention N will be manipulated using the standard powder: liquid ratio which is, one scoop of powder with one drop of liquid. Powder and liquid will be dispensed on the mixing pad and mixed using a plastic spatula according to the manufacturer's instruction for 45-60 seconds
  Arms: Cention N without adhesive.
Other: Cention N + Adhesive — Cavity will be rinsed with water to remove all residue. Etchant will be applied onto the prepared cavity for 15 seconds and thoroughly rinsed with water spray and gently dried with air jet. A layer of Tetric N Bond universal will be applied on the enamel & dentin surface using a disposable applicator, the material will be gently brushed into dentin for at least 10 seconds
  Arms: Cention N with adhesive
Other: Bulk Fill Composite — Cavity will be rinsed with water to remove all residue. Etchant will be applied onto the prepared cavity for 15 seconds and thoroughly rinsed with water spray and gently dried with air jet. A layer of Tetric N Bond universal will be applied on the enamel & dentin surface using a disposable applicator, the material will be gently brushed into dentin for at least 10 seconds.
  Arms: Filtek Bulk Fill posterior composite

SUMMARY:
Despite significant advances in composite materials, they are still perceived as technique-sensitive and exhibit failure related to excessive wear and polymerization shrinkage. Cention N is a recently introduced alkasite restorative that contains special reactive fillers. Its application in restorative dentistry may be significant, promoting remineralization of carious lesions & reduction of polymerization shrinkage. The study will aim to compare the clinical performance of Cention N (with and without adhesive) and composite resin (Filtek Bulk Fill) in class I restorations using FDI criteria. Thirty-six class I cavities will be selected and equally allocated into 3 groups: Group I (n=12): (Cention N with adhesive), Group II (n=12): (Cention N without adhesive) & Group III (n=12): composite resin (Filtek Bulk Fill) in class I cavities. Patients will be followed up at 1 week 3, 6, and 12 months and evaluated using the FDI criteria. Postoperative sensitivity, staining, and recurrent caries will be evaluated in this clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Permanent molars with occlusal pit and fissure caries.
* Good oral hygiene.
* Occlusal contact with antagonist teeth.

Exclusion Criteria:

* Permanent molars with occlusal pit and fissure caries.
* Good oral hygiene.
* Age between 18- 45 years.
* Occlusal contact with antagonist teeth.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2022-10-13 (Actual); Primary Completion 2023-11-28 (Actual); Study Completion 2023-11-28 (Actual)

PRIMARY OUTCOMES:
Change in pain sensitivity | 1 week, after 3, 6 and 12 months
  Air spray will be applied from a 2-mm distance on to the occlusal surface for 35seconds and should always be compared with the reaction of adjacent vital teeth. The severity of patients' pain/sensitivity will be recorded and given a score from 1 to 5
Change in occurrence of recurrent caries | 1 week, after 3, 6 and 12 months
  All surfaces were dried prior to evaluation. The restorations' assessment will be performed using a dental mirror and a ball-point probe aided by periapical radiographs.
Change in occurrence of marginal stains | 1 week, after 3, 6 and 12 months
  It is recommended to ask the patient about dietary habits. The restoration surface will be evaluated with regard to staining by comparison with the surrounding hard tissues and will be performed by the means of visual inspection aided with intraoral photography

CONTACTS AND LOCATIONS:
Locations (1):
- Alexandria Faculty of Dentistry, Alexandria, Egypt

REFERENCES:
- [Derived] El-Salamouny NA, Elmahy WA, Holiel AA. Comparative evaluation of bioactive alkasite-based material in different application modes: a 1-year randomized controlled clinical trial. Odontology. 2025 Oct;113(4):1689-1700. doi: 10.1007/s10266-025-01095-4. Epub 2025 Apr 15. PMID 40229532